CLINICAL TRIAL: NCT02668822
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Trial to Study the Efficacy and Safety of MK-8342B (ENG-E2 Vaginal Ring) in Women With Moderate to Severe Primary Dysmenorrhea
Brief Title: Efficacy and Safety of Etonogestrel + 17β-Estradiol Vaginal Ring (MK-8342B) in the Treatment of Women With Primary Dysmenorrhea (MK-8342B-060)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by Sponsor as a result of a business decision to discontinue the development program for MK-8342B for reasons unrelated to safety or efficacy.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8342B-060; 2015-004326-34 (EudraCT Number)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Endoglin; Contraceptive Devices, Female; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENG 125 μg + E2 300 μg (MK-8342B) (Experimental): Participants received up to 4 cycles of etonogestrel-17β estradiol (ENG-E2) at a daily dose of 125 μg/300 μg via vaginal ring. Each cycle consisted of 21 days of MK-8342B vaginal ring use followed by 7 ring-free days.
  Interventions: Drug: ENG 125 μg + E2 300 μg vaginal ring (MK-8342B); Drug: Ibuprofen
- Placebo (Placebo Comparator): Participants received up to 4 cycles of placebo via vaginal ring. Each cycle consisted of 21 days of placebo vaginal ring use followed by 7 ring-free days.
  Interventions: Drug: Placebo vaginal ring; Drug: Ibuprofen

INTERVENTIONS:
Drug: ENG 125 μg + E2 300 μg vaginal ring (MK-8342B) — Medicated vaginal ring
  Other Names: MK-8342B
  Arms: ENG 125 μg + E2 300 μg (MK-8342B)
Drug: Placebo vaginal ring — Placebo vaginal ring
  Arms: Placebo
Drug: Ibuprofen — Ibuprofen 400-mg tablets, to be taken orally, were provided to the participants for use as rescue medication for dysmenorrhea treatment throughout the study. Participants may have taken 400 mg every 4 hours as needed for pelvic pain/cramping.

SUMMARY:
The purpose of this study was to evaluate the efficacy of the etonogestrel (ENG) + 17β-estradiol (E2) (MK-8342B) vaginal ring compared to placebo vaginal ring in the treatment of dysmenorrhea at Treatment Cycle 2. This study was also to assess the safety and tolerability of the ENG-E2 vaginal rings over 4 treatment cycles. Primary hypothesis: Relative to the placebo ring, the ENG-E2 vaginal ring results in a greater proportion of participants with a ≥3-point reduction in peak pelvic pain score and no increase in the number of rescue pain relief (ibuprofen) tablets taken at Treatment Cycle 2 as compared to baseline.

DETAILED DESCRIPTION:
The cramping window for each participant was to be defined as a 4-day time interval that began the day prior to initiation of each cyclic bleeding episode (spontaneous menses or hormone withdrawal bleeding) and continued until the third bleeding day (inclusive). An external committee of blinded independent reviewers was to determine the 4-day cramping window for each participant so that analysis of the efficacy data could be conducted. The study was terminated early due to a business decision by the Sponsor to discontinue product development for reasons unrelated to safety or efficacy outcomes. Due to the early study termination, the blinded independent review committee that was supposed to determine the 4-day cramping windows for data analysis was not assembled; thus cramping windows were not determined. Without defined cramping windows, the efficacy outcome measures for this study could not be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarcheal female, age ≤50 years, in good physical and mental health.
* History of moderate to severe primary dysmenorrhea for the past 3 months or longer, and no history of recurrent non-menstrual pelvic pain intermittently or continuously throughout the month, and no history of dysmenorrhea secondary to structural pelvic pathology.
* Body mass index (BMI) of ≥18 and <38 kg/m^2.
* History of regular menstrual cycles with a cycle length between 24 and 32 days (inclusive) for the past three months.
* Willing to adhere to use of the vaginal ring and to all required trial procedures, and not planning to relocate during the study.
* Willing to use the rescue medication ibuprofen at the study recommended dose and no other pain medication for treatment of dysmenorrhea.

Exclusion Criteria:

* Cardiovascular risks and disorders, including history of venous thromboembolic [VTE] events, arterial thrombotic or thromboembolic [ATE] events, transient ischemic attack, angina pectoris, or claudication; at higher risk of VTE events due to recent prolonged immobilization, plans for surgery requiring prolonged immobilization, or a hereditary or acquired predisposition or elevated risk for venous or arterial thrombosis; currently smoking or uses tobacco/nicotine containing products and is ≥35 years of age; uncontrolled or severe hypertension; history of severe dyslipoproteinemia; <35 years of age with a history of migraine with aura or focal neurological symptoms or ≥35 years of age with a history of migraines with or without aura or focal neurologic symptoms; diabetes mellitus with end-organ involvement or >20 years duration; multiple cardiovascular risk factors such as ≥35 years of age, obesity, inadequately controlled hypertension, use of tobacco/ nicotine products, or inadequately controlled diabetes.
* Gynecologic conditions: surgically sterilized, has used hormonal contraceptives (pill, patch, ring, implant, intrauterine system) within the past 3 months, or currently uses non-hormonal intrauterine device (IUD); within past 6 months has had undiagnosed (unexplained) abnormal vaginal bleeding or any abnormal vaginal bleeding expected to recur during study; has gonorrhea, chlamydia, or trichomonas or symptomatic vaginitis/cervicitis; has abnormal cervical smear or positive high-risk human papillomavirus (HPV) test at screening or documented within 3 years of screening; has Stage 4 pelvic organ prolapse (1 cm beyond introitus) or lesser degrees of prolapse with history of difficulty retaining tampons, vaginal rings, or other products within vagina.
* Gastrointestinal and urologic disorders, including history of pancreatitis associated with severe hypertriglyceridemia; clinically significant liver disease, including active viral hepatitis or cirrhosis; or a history of the gastrointestinal or urologic tract which may cause pelvic pain.
* Other medical disorders, including history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer; any disease that may worsen under hormonal treatment such as disturbances in bile flow, systemic lupus erythematosus, pemphigoid gestationis or idiopathic icterus during previous pregnancy, middle-ear deafness, Sydenham chorea, or porphyria; known allergy/sensitivity or contraindication to the investigational products or their excipients; known allergy/sensitivity or contraindication to ibuprofen, or has experienced asthma, urticaria, or allergic-type reactions after taking aspirin, or other nonsteroidal anti-inflammatory drugs; history of drug or alcohol abuse or dependence.
* Known or suspected pregnancy, or had been pregnant or breastfeeding within past 2 months.
* Has used investigational drug and/or participated in other clinical trial within past 8 weeks.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ENG 125 μg + E2 300 μg (MK-8342B): Participants received up to 4 cycles of etonogestrel-17β-estradiol (ENG-E2) at a daily dose of 125 μg/300 μg via vaginal ring. Each cycle consisted of 21 days of MK-8342B vaginal ring use followed by 7 ring-free days.
Period: Overall Study
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Started | 9 | 9
Completed | 0 | 0
Not Completed | 9 | 9
Not completed — Protocol Violation | 2 | 0
Not completed — Study Terminated by Sponsor | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- ENG 125 μg + E2 300 μg (MK-8342B): Participants received up to 4 cycles of ENG-E2 at a daily dose of 125 μg/300 μg via vaginal ring. Each cycle consisted of 21 days of MK-8342B vaginal ring use followed by 7 ring-free days.
- Total: Total of all reporting groups
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (10) | 28 (5) | 30 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥3 Point Reduction in Peak Pelvic Pain Score and no Increase in Number of Ibuprofen Tablets Taken at Treatment Cycle 2, Compared to Baseline
Description: Participants were asked to rate their worst pain or cramps in the past 24 hours on a scale of 0 to 10 (0=No pain or cramps to 10=Extreme pain or cramps) and to indicate the number of ibuprofen tablets they took during the 4-day cramping window. The peak pelvic pain score was to be calculated as the highest (daily) pelvic pain score observed within the cramping window of the cycle and the total number of ibuprofen tablets taken was to be based on the 4-day cramping window. The baseline peak pelvic pain score and number of ibuprofen tablets taken were to be defined as the mean value of the 2 peak pelvic pain scores and the mean value of the total number of ibuprofen tablets taken during the cramping window of each of the 2 menstruations during the screening period, respectively. The percentage of participants with a reduction in peak pelvic pain score of ≥3 points and no increase in the use of ibuprofen at Treatment Cycle 2 as compared to baseline was to be presented.
Time Frame: Baseline 4-day cramping window and Treatment Cycle 2 4-day cramping window, as determined by committee for each participant
Population: The population was to consist of all participants in whom a vaginal ring was inserted & who had ≥1 day of diary entry each within a 4-day cramping window during a baseline cycle & a treatment cycle. Due to termination, the committee to determine cramping windows was not assembled, cramping windows were not determined & data could not be analyzed.
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 126 days
Population: The population consisted of all participants in whom a vaginal ring was inserted.
Measure: Number; unit: Participants
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 9 | 9
Participants | 0 | 1

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. The number of participants who discontinued study treatment due an AE is presented.
Time Frame: Up to approximately 112 days
Population: The population consisted of all participants in whom a vaginal ring was inserted.
Measure: Number; unit: Participants
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

4. Secondary Outcome: Change From Baseline in Peak Pelvic Pain Score at Treatment Cycle 2
Description: Participants were asked to rate their worst pain or cramps in the past 24 hours on a scale of 0 to 10 (0=No pain or cramps to 10=Extreme pain or cramps). The peak pelvic pain score was to be calculated as the highest (daily) pelvic pain score observed within the 4-day cramping window of the cycle. The baseline peak pelvic pain score was to be defined as the mean value of the 2 peak pelvic pain scores during the cramping window of each of the 2 menstruations during the screening period. The change from baseline in peak pelvic pain score at Treatment Cycle 2 was to be presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in the Number of Days With no Impact on Items of Physical, Work/School and Social/Leisure Activities at Treatment Cycle 2
Description: Participants were asked to indicate how much pain or cramps limited their physical, work/school and social/leisure activities and over the previous 24 hours. The level of negative impact of dysmenorrhea on daily life was scored on a 5-point scale (0=Not at all to 4=Extremely impacted). For each of the 3 impact items, the baseline score was to be defined as the mean value obtained from the 2 menstruations during the screening period. The change from baseline to Treatment Cycle 2 in the number of days during the cramping window with no impact of dysmenorrhea (score = 0) on each of the following items was to be presented: work/school, physical activities and leisure/social activities.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Pelvic Pain Score of "0" or "1" and no Use of Ibuprofen Tablets at Treatment Cycle 2
Description: Participants were asked to rate their worst pain or cramps on a scale of 0 to 10 (0=No pain or cramps to 10=Extreme pain or cramps) and to indicate the number of ibuprofen tablets they took during the 4-day cramping window. The percentage of participants with no or minimal pelvic pain (score of "0" or "1") and no use of ibuprofen at Treatment Cycle 2 was to be presented.
Time Frame: Treatment Cycle 2 4-day cramping window, as determined by committee for each participant
Population: The population was to consist of all participants in whom a vaginal ring was inserted & who had ≥1 day of diary entry each within a 4-day cramping window during Treatment Cycle 2. Due to termination, the committee to determine cramping windows was not assembled, cramping windows were not determined & data could not be analyzed.
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With ≥3-point Reduction in Peak Pelvic Pain Score and a Decrease in Number of Ibuprofen Tablets Taken at Treatment Cycle 2, Compared to Baseline
Description: Participants were asked to rate their worst pain or cramps in the past 24 hours on a scale of 0 to 10 (0=No pain or cramps to 10=Extreme pain or cramps) and to indicate the number of ibuprofen tablets they took during the 4-day cramping window. The baseline peak pelvic pain score and number of ibuprofen tablets taken were to be defined as the mean value of the 2 peak pelvic pain scores and the mean value of the total number of ibuprofen tablets taken during the cramping window of each of the 2 menstruations during the screening period, respectively. The percentage of participants with a reduction in peak pelvic pain score of ≥3 points and a decrease in the use of ibuprofen at Treatment Cycle 2 as compared to baseline was to be presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in the Mean Pelvic Pain Score at Treatment Cycle 2
Description: The mean pelvic pain score was to be calculated as the mean of the highest scores for pelvic pain observed within the 4-day cramping window of the screening or treatment cycle. The baseline mean pelvic pain score was to be defined as the mean value of the 2 mean pelvic pain scores of the 2 menstruations during the screening period. The change from baseline in mean pelvic pain score at Treatment Cycle 2 was to be presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study treatment (Up to approximately 126 days)
Description: The population consisted of all participants in whom a vaginal ring was inserted.
Arm/Group | ENG 125 μg + E2 300 μg (MK-8342B) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENG 125 μg + E2 300 μg (MK-8342B) (N=9) | Placebo (N=9)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.